CLINICAL TRIAL: NCT00803478
Title: The Effect of Hinge Position and Hinge Width on Corneal Sensation and Dry Eye After IntraLase LASIK Procedure
Acronym: IDES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shahzad Mian, erry J Bergstrom Collegiate Professor of Resident Education in Ophthalmology and Visual Sciences and Associate Professor of Oph, Ophthalmology & Visual Science, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM 18730-IDES
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Myopia
Keywords: IntraLase LASIK for primary myopia
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hinge position (Active Comparator): superior vs. temporal
  Interventions: Procedure: LASIK
- Hinge width (Active Comparator): 45 vs 90 degrees
  Interventions: Procedure: LASIK
- Flap Thickness (Active Comparator): 110 vs 130 microns
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: LASIK

SUMMARY:
Corneal sensation is known to play a role in tear secretion. Decreased sensation leads to decreased tear production; and when bilateral, leads to a decreased blink rate as well. Dry eyes are a common side effect of LASIK. Incidence rates vary widely, but have been reported in as many as 59% of patients. And almost all patients have some transient dry eye symptoms immediately following LASIK.

Previous studies have looked at the effect of hinge position (superior vs. nasal) and hinge width on corneal sensation and dry eye after LASIK performed with a mechanical microkeratome. Corneal sensation was decreased and dry eye signs and symptoms increased immediately following LASIK in all eyes. These parameters then improved at all time periods between 1 week and 6 months post-operative. Loss of corneal sensation and dry eye signs and symptoms were greater in eyes with superior-hinge flap than nasal-hinge flap, and in eyes with narrower hinge flap rather than wider hinge flap IntraLase LASIK, using the IntraLase femtosecond laser rather than a mechanical microkeratome to cut the corneal flap, has become an increasingly popular procedure. It provides several advantages over mechanical microkeratomes, including reduced surgical complications, more predictable flap thickness, better astigmatic neutrality, decreased epithelial injury, and an ability to operate on a wider range of patients.

The investigators propose this study to evaluate the effect of flap hinge size and flap thickness in corneal flaps created with the IntraLase laser. The investigators would like to determine if there is a difference from the previously discussed results found when using the mechanical microkeratome. Also, with the increased ease of programming alternate hinge width or flap thickness with IntraLase, if the investigators find a significant difference with an alternate flap configuration, it might translate to a feasible change in clinical practice.

DETAILED DESCRIPTION:
Corneal innervation/sensation is supplied by the long ciliary nerves which branch from the trigeminal nerve. The nerves enter the cornea in the mid-stroma at the nasal and temporal limbus. They then branch and turn anterior to form a dense plexus sub-Bowman's layer. The nerves finally terminate in the wing cell layer from where they enervate the epithelium. Corneal sensation has been shown to be decreased after all corneal surgeries, including LASIK.

Corneal sensation is known to play a role in tear secretion. Decreased sensation leads to decreased tear production; and when bilateral, leads to a decreased blink rate as well. Dry eyes are a common side effect of LASIK. Incidence rates vary widely, but have been reported in as many as 59% of patients. And almost all patients have some transient dry eye symptoms immediately following LASIK.

Previous studies have looked at the effect of hinge position (superior vs. nasal) and hinge width on corneal sensation and dry eye after LASIK performed with a mechanical microkeratome.1,2 Corneal sensation was decreased and dry eye signs and symptoms increased immediately following LASIK in all eyes. These parameters then improved at all time periods between 1 week and 6 months post-operative. Loss of corneal sensation and dry eye signs and symptoms were greater in eyes with superior-hinge flap than nasal-hinge flap, and in eyes with narrower hinge flap rather than wider hinge flap IntraLase LASIK, using the IntraLase femtosecond laser rather than a mechanical microkeratome to cut the corneal flap, has become an increasingly popular procedure. It provides several advantages over mechanical microkeratomes, including reduced surgical complications, more predictable flap thickness, better astigmatic neutrality, decreased epithelial injury,3 and an ability to operate on a wider range of patients.

We propose this study to evaluate the effect of flap hinge position and size in corneal flaps created with the IntraLase laser. We would like to determine if there is a difference from the previously discussed results found when using the mechanical microkeratome. Also, with the increased ease of programming alternate hinge position and width with IntraLase, if we find a significant difference with an alternate flap configuration, it might translate to a feasible change in clinical practice.

Specific Aims: To evaluate the effect of hinge position (superior vs. temporal) , hinge width (45 vs. 90 degrees), and flap thickness on corneal sensation and dry eye after IntraLase LASIK.

ELIGIBILITY:
Inclusion Criteria:

* Refractive error: Myopia < 12 D, with astigmatism < 3 D,
* Age > 20 y/o
* Regular corneal curvature, sufficient corneal thickness, appropriate pupil size, normal slit lamp examination
* Informed consent to permit us to use their records for this study without using name, medical record number, or date of surgery.

Exclusion Criteria:

* Pregnant/nursing
* Systemic collagen vascular disease
* Autoimmune disease
* Severe dry eyes

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-06; Primary Completion 2008-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of hinge position (superior vs. temporal) , hinge width (45 vs. 90 degrees), and flap thickness on corneal sensation and dry eye after IntraLase LASIK. | pre operative and 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Cornea Clinic, Kellogg Eye Center, Ann Arbor, Michigan, United States